CLINICAL TRIAL: NCT02061423
Title: Pilot Phase I HER-2 Pulsed DC Vaccine to Prevent Recurrence for Patients With HER-2 Driven High Risk Invasive Breast Cancer Post Neoadjuvant Chemotherapy
Brief Title: HER-2 Pulsed DC Vaccine to Prevent Recurrence of Invasive Breast Cancer Post Neoadjuvant Chemotherapy
Acronym: Neoadjuvant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-18776; UPCC26113 (Other: CTSRMC, Abramson Cancer Center, University of Pennsylvania); NCT02110199 (obsolete NCT alias)
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: Invasive Breast Cancer; Breast Cancer; Immunotherapy; Vaccine; Dendritic Cell; Neoadjuvant
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HER-2 Pulsed Dendritic Cell Vaccine (Experimental): 6 weekly HER-2 pulsed dendritic cell vaccines followed by 3 booster vaccines once every 3 months.
  Interventions: Biological: HER-2 pulsed Dendritic Cell Vaccine

INTERVENTIONS:
Biological: HER-2 pulsed Dendritic Cell Vaccine — Each dose will consist of between 1.0-2.0 x 10^7 cells and will be injected into 1-2 different normal groin lymph nodes or axillary nodes.

SUMMARY:
The primary goals of this trial will be to determine the safety and immune activity of HER-2 pulsed DC1 vaccine in patients with high risk HER-2pos breast cancer with residual disease post neoadjuvant therapy. Investigators will also explore the possibility of determining whether circulating tumor cells can be used as surrogate to assess response to vaccination.

DETAILED DESCRIPTION:
Dendritic cell cancer vaccines combined with chemotherapy may increase complete responses giving breast cancer specific immune cells greater opportunity to function while the immune repertoire is being shifted by chemotherapy to anti-breast cancer response and offer the chance to test secondary prevention of breast cancer in high risk settings. There is a need to determine whether this ICAIT DC1 can activate CD4 and CD8 T cells prior to or in combination with chemotherapy with or without added trastuzumab.

This study began at the Abramson Cancer Center of the University of Pennsylvania and will be continued at H. Lee Moffitt Cancer Center and Research Institute.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years.
* HER-2 expressing stage I - III breast cancer with residual disease in the breast or axillary nodes post-neoadjuvant chemotherapy.
* Women of childbearing age with a negative pregnancy serum test documented prior to enrollment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status Score of 0 or 1.
* Women of childbearing potential must agree to use a medically acceptable form of birth control during their participation in the study.
* Have voluntarily signed a written Informed Consent in accordance with institutional policies after its contents have been fully explained to them.

Exclusion Criteria:

* Pregnant or lactating.
* Positive for HIV or hepatitis C at baseline by self report.
* Potential participants with coagulopathies, including thrombocytopenia with platelet count <75,000, INR > 1.5 and partial thromboplastin time > 50 sec.
* Potential participants with MUGA < 50% EF.
* Pre-existing medical illnesses or medications which might interfere with the study as determined by Principal Investigator (PI).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-04-08 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Participation Compliance | Up to 18 months
  Feasibility: Defined as a patient's ability and willingness to complete the treatment regimen (6 weekly vaccinations). Data collection will include rate of successful completion and occurrence rate for each reason stated for non-completion.
Occurrence of Treatment Related Adverse Events | Up to 18 months
  Number of participants with treatment related adverse events, per event category.

SECONDARY OUTCOMES:
Immunogenicity | Up to 5 years follow-up
  Immunogenicity will be evaluated by descriptive statistics, plots of pre- and post-treatment values and fold changes. Immune response rate and 95% exact confidence interval will be calculated.
Anti-HER2 Immunity | Up to 5 years follow-up
  Anti-HER2 response will be quantitated as EOS/baseline fold change in dilution studies.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Czerniecki, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Czerniecki BJ, Roses RE, Koski GK. Development of vaccines for high-risk ductal carcinoma in situ of the breast. Cancer Res. 2007 Jul 15;67(14):6531-4. doi: 10.1158/0008-5472.CAN-07-0878. PMID 17638860
- [Background] Czerniecki BJ, Koski GK, Koldovsky U, Xu S, Cohen PA, Mick R, Nisenbaum H, Pasha T, Xu M, Fox KR, Weinstein S, Orel SG, Vonderheide R, Coukos G, DeMichele A, Araujo L, Spitz FR, Rosen M, Levine BL, June C, Zhang PJ. Targeting HER-2/neu in early breast cancer development using dendritic cells with staged interleukin-12 burst secretion. Cancer Res. 2007 Feb 15;67(4):1842-52. doi: 10.1158/0008-5472.CAN-06-4038. Epub 2007 Feb 9. PMID 17293384
- [Background] Koski GK, Koldovsky U, Xu S, Mick R, Sharma A, Fitzpatrick E, Weinstein S, Nisenbaum H, Levine BL, Fox K, Zhang P, Czerniecki BJ. A novel dendritic cell-based immunization approach for the induction of durable Th1-polarized anti-HER-2/neu responses in women with early breast cancer. J Immunother. 2012 Jan;35(1):54-65. doi: 10.1097/CJI.0b013e318235f512. PMID 22130160
- [Background] Sharma A, Koldovsky U, Xu S, Mick R, Roses R, Fitzpatrick E, Weinstein S, Nisenbaum H, Levine BL, Fox K, Zhang P, Koski G, Czerniecki BJ. HER-2 pulsed dendritic cell vaccine can eliminate HER-2 expression and impact ductal carcinoma in situ. Cancer. 2012 Sep 1;118(17):4354-62. doi: 10.1002/cncr.26734. Epub 2012 Jan 17. PMID 22252842
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/